CLINICAL TRIAL: NCT03051659
Title: A Randomized Phase II Study Of Eribulin Mesylate With Or Without Pembrolizumab For Metastatic Hormone Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigaor, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-577
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eribulin Mesylate (Experimental): -Eribulin mesylate will be administered on Days 1 and 8 of each 21 day cycle for 1.4mg/m^2 intravenously.
  Interventions: Drug: Eribulin Mesylate
- Eribulin Mesylate Combine with Pembrolizumab (Experimental): * Pembrolizumab will be administered in clinic once per cycle, given 200mg/m^2 intravenously prior to Eribulin Mesylate.
  * Eribulin mesylate will be administered on Days 1 and 8 of each 21 day cycle for 1.4 mg/m^2 intravenously.
  Interventions: Drug: Eribulin Mesylate; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate is developed from a natural substance found in a sea sponge. Eribulin mesylate works by preventing cancer cells from multiplying
  Other Names: Halaven
Drug: Pembrolizumab — Pembrolizumab binds to PD-1, an inhibitory signaling receptor expressed on the surface of activated T cells, and blocks the binding to and activation of PD-1 by its ligands, which results in the activation of T-cell-mediated immune responses against tumor cells.
  Other Names: Keytruda
  Arms: Eribulin Mesylate Combine with Pembrolizumab

SUMMARY:
This research study is exploring chemotherapy in combination with immunotherapy (a therapy that uses the body's own immune system to control cancer) as a possible treatment for metastatic hormone receptor positive breast cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

In this research study, The investigators are evaluating the safety and effectiveness of Eribulin mesylate with or without Pembrolizumab in metastatic hormone receptor positive breast cancer.

The FDA (the U.S. Food and Drug Administration) has not approved the combination of Pembrolizumab and Eribulin mesylate for Breast Cancer.

The FDA has not approved Pembrolizumab for this specific type of breast cancer but it has been approved in the United States for other diseases.

The FDA has approved Eribulin mesylate as a treatment option for this type of breast cancer.

Pembrolizumab is a medicine that may treat cancer by working with the immune system. The immune system is the body's natural defense against disease. The immune system sends types of cells called "T cells" throughout the body to detect and fight infections and diseases, including cancer. For some types of cancer, the T cells do not work as they should and are prevented from attacking the tumors. Pembrolizumab is thought to work by blocking a protein in the T cells called PD-1 ("programmed death 1"), which then may allow these cells and other parts of the immune system to attack tumors.

Eribulin mesylate is developed from a natural substance found in a sea sponge. Eribulin mesylate works by preventing cancer cells from multiplying.

The combination of Pembrolizumab and Eribulin mesylate is investigational. The study drugs, when given separately, work in different ways to stop the cancer cells from growing and spreading. However, it is not known if giving the two study drugs at the same time will have a better anti-cancer effect than giving each treatment on its own.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically or cytologically confirmed Stage IV invasive breast cancer. Patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Subjects must have at least one lesion that is not within a previously radiated field that is evaluable on computerized tomography (CT) or magnetic resonance imaging (MRI) scan per RECIST version 1.1. If the subject's only evaluable disease is within a previously radiated field, it must have demonstrated progression since the time of radiation.
* Participants must have HR positive, HER2-negative breast cancer (ER>1% and/or, PR>1%, HER2-negative per ASCO CAP guidelines, 2013 resulted on the primary tumor and/or a metastatic lesion).
* Participants must have already received or been intolerant to at least two lines of hormonal therapies (including the adjuvant or metastatic setting) or be appropriate candidates for chemotherapy
* Prior chemotherapy: Participants are allowed to have received up to 2 prior lines of chemotherapy in the metastatic setting. If a prior chemotherapy was given for less than 1 cycle, it will not be counted as a prior line. The last dose of chemotherapy must be ≥14 days prior to initiation of study therapy. Participants should be adequately recovered from acute toxicities of prior treatment. No prior treatment with eribulin mesylate is allowed.
* Prior biologic therapy: The last dose of biologic or investigational therapy must be ≥21 days prior to initiation of study therapy.
* Prior hormonal therapy: Hormonal therapy must have been discontinued ≥14 days prior to initiation of study therapy. However, continuation of ovarian suppression is allowed.
* Prior radiation therapy: Participants may have received prior radiation therapy in either the metastatic or early-stage setting. Radiation therapy must be completed ≥14 days prior to initiation of study therapy.
* Prior targeted therapy: Targeted therapy must have been discontinued ≥ 14 days prior to initiation of study therapy.
* Biphosphonates/Denosumab: Participants on bisphosphonates/denosumab may continue receiving bisphosphonate therapy during study treatment.
* Participants must have an archival tumor sample available (1 block or 20 unstained slides). If no archival tissue is available, participants must be willing to undergo a research biopsy of their disease if it is safely accessible.
* Age ≥ 18 years of age
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Participants must have normal organ and marrow function as defined below:
* absolute neutrophil count ≥1,500/mcL
* platelets ≥100,000/mcL
* hemoglobin ≥ 8 g/dl
* total bilirubin ≤1.5 × institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN (≤ 5 × institutional ULN with documented liver metastases,
* serum creatinine ≤1.5mg/dL or calculated GFR ≥60 mL/min
* INR/PT ≤1.5 times ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* aPTT/PTT ≤1.5 times ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* The effects of eribulin mesylate and pembrolizumab on the developing human fetus are unknown. Pre-clinical data was suggestive of a teratogenic effect of eribulin mesylate. For these reasons women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and 4 months after the last dose of eribulin mesylate and/or pembrolizumab. Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the treating physician and principal investigator should be informed immediately.
  * While on the study, women must not breastfeed.
  * Subjects of childbearing potential are defined as those who have not been surgically sterilized and/or have had a menstrual period in the past year
* Female subjects of childbearing potential, as defined above, must have a either a negative urine or a negative serum pregnancy test within seven (7) days of first dose of pembrolizumab. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria

* Chemotherapy-related or radiation-related toxicities that have not resolved to Grade 1 severity or lower, except for stable sensory neuropathy (≤ Grade 2) and alopecia.
* Participants who are receiving any other investigational agents.
* Previous treatment with eribulin mesylate or any anti-PD-1, PD-L1, or PD-L2 agent or participation in any MK-3475 Merck studies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to eribulin mesylate or pembrolizumab.
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with previously diagnosed brain metastases are eligible if they have completed treatment at least 4 weeks prior to registration, are neurologically stable and absence of new neurologic symptoms for the last 4 weeks prior to study entry, and have recovered from the effects of radiotherapy or surgery. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥2 weeks before the first study drug. Treatment for brain metastases may have included whole brain radiotherapy, radiosurgery, or a combination as deemed appropriate by the treating physician.
* Uncontrolled intercurrent illness, including, but not limited to uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure-New York Heart Association Class III or IV, active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, gastric or duodenal ulceration diagnosed within the previous 6 months, chronic liver or renal disease, severe malnutrition or psychiatric illness/social situations that would limit compliance with study requirements.
* Clinically significant electrocardiogram (ECG) abnormality, including a marked baseline prolonged QT/QTc ([QT interval/corrected QT interval], eg, a repeated demonstration of a QTc interval >500 ms).
* Medcial condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. For example, participants with autoimmune disease that requires systemic steroids or immunosuppression agents should be excluded. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History or evidence of active, noninfectious pneumonitis that required treatment with steroids.
* History of interstitial lung disease.
* Participants known to be positive for the human immunodeficiency virus (HIV), Hepatitis B antigen (HepBsAg), or Hepatitis C virus (HCV) RNA. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Pembrolizumab and/or eribulin mesylate. In addition, these participants are at increased risk of lethal infections.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 5 years and felt to be at low risk of recurrence should be discussed with the study sponsor to determine eligibility.
* Has received a live vaccine within 28 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keenan TE, Guerriero JL, Barroso-Sousa R, Li T, O'Meara T, Giobbie-Hurder A, Tayob N, Hu J, Severgnini M, Agudo J, Vaz-Luis I, Anderson L, Attaya V, Park J, Conway J, He MX, Reardon B, Shannon E, Wulf G, Spring LM, Jeselsohn R, Krop I, Lin NU, Partridge A, Winer EP, Mittendorf EA, Liu D, Van Allen EM, Tolaney SM. Molecular correlates of response to eribulin and pembrolizumab in hormone receptor-positive metastatic breast cancer. Nat Commun. 2021 Sep 21;12(1):5563. doi: 10.1038/s41467-021-25769-z. PMID 34548479
- [Derived] Tolaney SM, Barroso-Sousa R, Keenan T, Li T, Trippa L, Vaz-Luis I, Wulf G, Spring L, Sinclair NF, Andrews C, Pittenger J, Richardson ET 3rd, Dillon D, Lin NU, Overmoyer B, Partridge AH, Van Allen E, Mittendorf EA, Winer EP, Krop IE. Effect of Eribulin With or Without Pembrolizumab on Progression-Free Survival for Patients With Hormone Receptor-Positive, ERBB2-Negative Metastatic Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1598-1605. doi: 10.1001/jamaoncol.2020.3524. PMID 32880602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from April 6, 2017, through August 28, 2018.
Period: Treatment Period
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Started | 44 | 46
Completed | 44 | 44
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Survival Follow-up
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Started | 44 | 44
Completed | 21 | 22
Not Completed | 23 | 22
Not completed — Lost to Follow-up | 23 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Customized [Median (Full Range); unit: years] | 57 [37 to 76] | 58 [30 to 76] | 57 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 87
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 41 | 81
  Asian | 2 | 0 | 2
  Black/African American | 0 | 2 | 2
  Other/Multiple | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease assessments is performed every 3 cycles (3 weeks/cycle) for the first 18 cycles. Median follow-up 10.5 months with range 0.43-19 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Number analyzed (Participants) | 22 | 21
months | 4.2 [3.7 to 6.1] | 4.1 [3.5 to 6.2]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response rate (ORR) was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease assessments is performed every 3 cycles (3 weeks/cycle) for the first 18 cycles. If after Cycle 18 scans, a participant has SD or better by RECIST the frequency of assessments may be reduced to every 4 cycles, up to a maximum of 18 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Number analyzed (Participants) | 44 | 44
percentage of participants | 34 [20.5 to 49.9] | 27 [14.9 to 42.8]

3. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive. Patients who discontinued treatment to pursue potentially curative resection were censored for progression-free survival at the time of surgery. Patients who had not experienced cancer progression or died were censored at their last known follow-up date.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Number analyzed (Participants) | 44 | 44
months | 12.5 [8.6 to NA] — insufficient number of participants with events | 13.4 [10.4 to NA] — insufficient number of participants with events

4. Secondary Outcome: Median Duration of Response (DOR)
Description: DOR is defined as the time from CR or PR achieved until renewed disease progression is detected. DOR will be calculated per RECIST 1.1 and irRECIST criteria.
Time Frame: Disease assessments is performed every 3 cycles (3 weeks/cycle) for the first 18 cycles. If after Cycle 18 scans, a participant has SD or better by RECIST the frequency of assessments may be reduced to every 4 cycles.
Measure: Median (Full Range); unit: months
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Number analyzed (Participants) | 44 | 44
months | 2.1 [1.0 to 4.6] | 0.6 [0 to 1.0]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Number analyzed (Participants) | 44 | 44
Participants | 21 | 22

6. Secondary Outcome: Number of Participants With Grade 3 or Higher Treatment-Related Toxicity
Description: All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate | Eribulin Mesylate Combine With Pembrolizumab
Number analyzed (Participants) | 44 | 44
Participants | 44 | 44

ADVERSE EVENTS:
Time Frame: Disease assessments is performed every 3 cycles (3 weeks/cycle) for the first 18 cycles. If after Cycle 18 scans, a participant has SD or better by RECIST the frequency of assessments may be reduced to every 4 cycles, up to a maximum of 18 months.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Arm/Group | Eribulin Mesylate Combine With Pembrolizumab | Eribulin Mesylate
All-Cause Mortality (participants affected / at risk) | 19/44 | 21/44
Serious Adverse Events (participants affected / at risk) | 27/44 | 25/44
Other Adverse Events (participants affected / at risk) | 44/44 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate Combine With Pembrolizumab (N=44) | Eribulin Mesylate (N=44)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 4
Alkaline phosphatase increased (Investigations) | 0 | 3
Anemia (Blood and lymphatic system disorders) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 4
Blood bilirubin increased (Investigations) | 1 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Investigations - Other, specify (Investigations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 16 | 16
Pain (General disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 3
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
White blood cell decreased (Investigations) | 3 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate Combine With Pembrolizumab (N=44) | Eribulin Mesylate (N=44)
Abdominal pain (Gastrointestinal disorders) | 8 | 6
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 17 | 14
Alkaline phosphatase increased (Investigations) | 11 | 9
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 19
Anemia (Blood and lymphatic system disorders) | 14 | 14
Anorexia (Metabolism and nutrition disorders) | 18 | 19
Anxiety (Psychiatric disorders) | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8
Ascites (Gastrointestinal disorders) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 24 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Blood bilirubin increased (Investigations) | 6 | 4
Blurred vision (Eye disorders) | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Breast pain (Reproductive system and breast disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Cardiac troponin T increased (Investigations) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 4 | 6
Cholesterol high (Investigations) | 2 | 0
Constipation (Gastrointestinal disorders) | 16 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 7
Creatinine increased (Investigations) | 4 | 1
Death NOS (General disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Depression (Psychiatric disorders) | 6 | 3
Diarrhea (Gastrointestinal disorders) | 18 | 12
Dizziness (Nervous system disorders) | 9 | 5
Dry mouth (Gastrointestinal disorders) | 5 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 7 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Edema limbs (General disorders) | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 2 | 0
Eye infection (Infections and infestations) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 39 | 39
Fever (General disorders) | 9 | 13
Flatulence (Gastrointestinal disorders) | 1 | 0
Flu like symptoms (General disorders) | 6 | 8
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gait disturbance (General disorders) | 1 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 3 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 8
Growth suppression (Musculoskeletal and connective tissue disorders) | 0 | 1
Gum infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 13 | 12
Hematuria (Renal and urinary disorders) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 6 | 5
Hyperthyroidism (Endocrine disorders) | 6 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 7 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 3
Hypotension (Vascular disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 8 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 2 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 5
Irritability (General disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Localized edema (General disorders) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphedema (Vascular disorders) | 1 | 2
Lymphocyte count decreased (Investigations) | 3 | 4
Mucosal infection (Infections and infestations) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 9 | 8
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 6 | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Nausea (Gastrointestinal disorders) | 25 | 28
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 3
Neutrophil count decreased (Investigations) | 17 | 23
Non-cardiac chest pain (General disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 20 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 24 | 26
Photophobia (Eye disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 6
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 3
Thromboembolic event (Vascular disorders) | 3 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper respiratory infection (Infections and infestations) | 1 | 2
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 1
Vaginal dryness (Reproductive system and breast disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 15 | 9
Watering eyes (Eye disorders) | 2 | 3
Weight loss (Investigations) | 7 | 3
White blood cell decreased (Investigations) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT03051659/Prot_SAP_000.pdf